CLINICAL TRIAL: NCT02042105
Title: A Prospective Epidemiologic and Clinical Feature Study of Non-Small Cell Lung Cancer (NSCLC) Patients With ALK Positive in China
Brief Title: A Prospective Epidemiologic Study of ALK-Positive NSCLC in China
Acronym: C-TALK
Status: Completed | Type: Observational
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG1303
Record Dates: First submitted 2013-11-09; First posted 2014-01-22 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Non-small-cell Lung Cancer
Keywords: non-small-cell lung cancer; anaplastic lymphoma kinase; immunohistochemistry
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a post-marketing, observational, non-interventional, multi-central study of patients with non-small cell lung cancer (NSCLC), with data collected prospectively from medical records at inclusion. The primary objective is to obtain the epidemiologic data of anaplastic lymphoma kinase (ALK)-positive in unselected Chinese patients with NSCLC.

DETAILED DESCRIPTION:
Archived paraffin-embedded and fresh frozen NSCLC tumor tissue will be obtained via the Department of Pathology. ALK positive status will be detected by Ventana immunohistochemistry (IHC) (Ventana Medical Systems, Inc. and Roche Diagnostics International, Inc). When ALK positive patients are detected, crizotinib will be administrated by various solutions based on physician's desecration and patients' willingness.

The secondary objectives include: 1.To obtain the epidemiologic data of ALK positive in unselected Chinese patients with NSCLC.2.To describe demographic, socioeconomic [such as age, gender, race/ethnicity, geographic location (including rural/urban area), pathologic parameters, education, family income, National Reimbursement Drug List (NRDL) or Provincial Reimbursement List (PRDL)], and clinical characteristics of NSCLC patients with ALK positive.

The exploratory objective is to describe prognosis patterns associated with crizotinib treated patients when efficacy data are available non-interventionally.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years), both sex.
* Histologically or cytologically proven diagnosis of primary NSCLC, including squamous cell carcinoma and adenocarcinoma.
* Written informed consent.

Exclusion Criteria:

* Those lung cancers without pathological diagnosis should not be included in case of other types of cancer, including small cell lung cancer (SCLC) or metastatic disease from other organs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unselected Chinese patients with non-small-cell lung cancer
Sampling Method: Probability Sample
Enrollment: 3649 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2016-07-06 (Actual)

PRIMARY OUTCOMES:
the frequency of ALK rearrangement in unselected Chinese patients with non-small cell lung cancer | one and half years

SECONDARY OUTCOMES:
demographic, socioeconomic,clinical and pathological features of ALK-positive NSCLC patients | one and half years

OTHER OUTCOMES:
prognosis patterns associated with crizotinib treated patients when efficacy data are available non-interventionally. | one and half years

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, MD, Principal Investigator — Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences; Yi-Long Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (2):
- China (2):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong